CLINICAL TRIAL: NCT06493097
Title: Hypnotherapy With Audiofiles for Children and Adolescents With Disorders of Gut-brain Interactions in Sweden -a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ola Olen, associate professor, senior consultant i pediatric gastroenterology, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00296-01
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Self-hypnosis; Functional Bowel Disorder; Functional Abdominal Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with hypnotherapy audio files (Experimental): Participants get access to a website, where they can find information about the diagnosis DGBI and mechanisms leading to symtoms. On the website they also get access to a tretament protocoll for self-hypnosis with audio files (5 different audio files, age-adjusted). Participants listen to audio files min 5 times/week for 12 weeks. They answer the study questionnaries before, after and every 3 weeks during the treatment.
  Interventions: Behavioral: Gut-directed hypnotherapy via audio files

INTERVENTIONS:
Behavioral: Gut-directed hypnotherapy via audio files — 5 audio files 10-15 min each, min 5 times a week for 12 weeks

SUMMARY:
This study aims at testing the effect and feasibility of a new treatment strategy - hypnotherapy mediated with audio files - for children and adolescents with disorders of gut-brain-interaction (DGBI) in Sweden. The treatment protocol has been used and studied in Netherlands, but the investigators have translated and formed it to suit the Swedish population. This study is a feasibility study that is followed by a large RCT to compare different psychological treatment options for this patient group.

If hypnotherapy mediated via audio files proves to be effective and feasible for this patient group, it would mean:

1. An exponential increase in the availability of evidence-based treatments. The hypnotherapy treatment is markedly easier to distribute than e.g. cognitive behavior therapy (CBT) which requires chat contact with a psychologist and is made available regardless of where in Sweden the family lives. In addition to shortened waiting times for patients, this would decrease the pressure in somatic care.
2. Possibility to offer tailored treatments. No treatment works for everyone. It is reasonable to assume that treatments with such different focuses as hypnotherapy and exposure-based CBT may be differently effective for different patients. A new treatment option can help a larger proportion of patients.
3. A more cost-effective treatment. Gut-directed hypnotherapy with audio files is a very inexpensive treatment, which would likely result in significant cost savings for this patient population.

DETAILED DESCRIPTION:
Hypnotherapy has shown promising results in international studies for treatment of DGBI. Gut-directed hypnotherapy for children is based on relaxation and imagery and sensation exercises with a focus on gastrointestinal symptoms ("directed daydreams", which both divert and provide a pleasant feeling in the body, which the child can use when the symptoms come). The aim is to both improve awareness of and increase control over the symptoms. Hypnotherapy is a safe treatment that has been shown to have minimal side effects. The research group in the Netherlands with whom investigators collaborate in this project has shown a significantly better effect in short and long term with hypnotherapy than with conventional medical treatment for children and adolescents with DGBI. Hypnotherapy via home-based self-exercises with audio files is proven as effective as individual therapy performed face-to-face by a therapist.

Preliminary results/ backround work: Collaboration with the Dutch group started, the treatment manual for gut-directed hypnotherapy has been translated into Swedish and has undergone cultural validation by experienced child psychologists and has been recorded in audiobook quality. The study website (where the families have access to the treatments and measure the outcomes) has been created. Comprehensive patient information material has been created about DGBI and hypnotherapy, which consists of both texts, films, and audio to reach all patient types (Fig 1a-b). The pilot study is ongoing since Sep 2023.

Aim: To test the practical aspects concerning patient recruitment, information about treatment, the treatment itself, measurement of outcome, required power for the main outcome. The lessons learned will help investigators to fine-tune the protocol and give the planned large RCT optimal conditions.

Study population: 30 patients (8-17 years, of which approximately half are 13-17 years) from Sachsska Children's Hospital's Gastrointestinal Clinic and Pediatric and Adolescent Medical Clinics in Stockholm, who are diagnosed with DGBI following Rome IV criteria. Before inclusion, the families meet with a study physician and a study nurse for an assessment of inclusion and exclusion criteria, for information about the study, and review of treatment principles.

Exposure: Gut-directed hypnotherapy exercises 5 times/week, for 12 weeks, delivered via audio files on the study's website (files can also be downloaded to mobile phone).

Outcome: At the beginning and end of the treatment and every third week during the treatment, the patients and parents will fill in self-assessments in the form of internationally validated questionnaires for symptom severity, quality of life, school absence etc, via an internet platform with identification control (which we have worked with in many previous projects). Improvement by >30% on the primary outcome measure is defined as clinically significant, based on international recommendations.

Power: In several previous pilot studies, 30 patients have been sufficient to obtain meaningfully tight confidence intervals for the outcome measures and to be able to conclude for future RCTs. However, no formal power analysis is relevant without a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: irritable bowel syndrome, functional abdominal pain, functional dyspepsia (following the Rome IV diagnostic criteria)
* The participant and at least one of the parents must understand Swedish

Exclusion Criteria:

* other medical condition that better explains the symtoms
* Absence from school >40% and/or psychiatric diagnosis that is judged to be more primary than the gastrointestinal problems, in these cases the children/young people are judged to need more intensive and multi-professional treatment

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ola Olén, MD PhD prof, Principal Investigator — Department of clinical epidemiology, Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children and adolescents with DGBI aged 8-17 years at the start of the treatment were recruited from Sachs Children's Hospital and four outpatient pediatric clinics in Stockholm between October 2023 and June 2024.
Pre-assignment Details: Participants received the intervention within 4 weeks from enrollment, all participants received same intervention in this pilot study.
Groups:
- Treatment With Hypnotherapy Audio Files: Participants get access to a website, where they can find information about the diagnosis DGBI and mechanisms leading to symtoms. On the website they also get access to a tretament protocoll for self-hypnosis with audio files (5 different audio files, age-adjusted). Participants listen to audio files min 5 times/week for 12 weeks. They answer the study questionnaries before and after the treatment.
Period: Overall Study
Arm/Group | Treatment With Hypnotherapy Audio Files
Started | 32
Completed | 25
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Sweden | 32
Symtom duration >2 years [Count of Participants; unit: Participants] | 24
Diagnosis IBS (irritable bowel syndrome) [Count of Participants; unit: Participants] | 22
Diagnosis FAP-NOS (functional abdominal pain - not otherwise specified) [Count of Participants; unit: Participants] | 5
Diagnosis FD (functional dyspepsia) [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Secondary Outcome: Pain Frequency and Intensity
Description: FACES pain scale. Minimum value 0, maximum value 10, higher score means worse outcome.
Time Frame: Week 0 (pre) and 12 (post) of treatment. The post-treatment measurement must be finished within 2 weeks from end of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale
  Baseline | 5.69 (2.28)
  Post-intervention | 4.54 (2.3)

2. Secondary Outcome: Stress
Description: PAS pediatric stress questionnare. Minimum value 0, maximum value 44, higher score means worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale
  Baseline | 15.78 (10.33)
  Post-intervention | 19.4 (11.15)

3. Secondary Outcome: Gastrointestinal Symtom -Related Anxiety
Description: BRQ-C questionnare. Minimum value 11, maximum value 77, higher score means worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale
  Baseline | 35.59 (13.38)
  Post-intervention | 35.65 (13.64)

4. Secondary Outcome: GI Symptom Specific Anxiety
Description: Visceral sensitivity index short scale. Minimum value 0, maximum value 35, higher score means worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale
  Baseline | 17.38 (9.14)
  Post-intervention | 6.56 (8.22)

5. Secondary Outcome: Quality of Life
Description: Peds-QL- QOL. Minimum value 0, maximum value 100, higher score means better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale
  Baseline | 70.48 (11.68)
  Post-intervention | 73.54 (15.59)

6. Secondary Outcome: Adequate Relief
Description: SAQ. Minimum value 0, maximum value 7, higher score means better outcome.
Time Frame: Week 12 (post) treatment. The post-treatment measurement must be finished within 2 weeks from end of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale | 4.12 (0.83)

7. Primary Outcome: Peds-QL-gastro
Description: Short questionnaire gastrointestinal symptom scale. Minimum value 0, maximum value 100, higher score means better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Hypnotherapy Audio Files
Number analyzed (Participants) | 25
units on a scale
  Baseline | 49.91 (13.43)
  Post-intervention | 60.15 (14.01)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow up, up to 12 weeks
Description: Hypnotherapy with audio files is considered a safe intervention that has no reported adverse effects in previous studies. The participants were instructed to self-report possible side effects in this study.
Arm/Group | Treatment With Hypnotherapy Audio Files
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
The within-group study design is a limitation, as true efficacy cannot be assessed while regression toward the mean cannot be controlled for. Another limitation was the lack of reliable compliance reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT06493097/Prot_SAP_000.pdf